CLINICAL TRIAL: NCT06354400
Title: The Effect of Core Stabilization Training on Chest Expansion, Functional Capacity, and Trunk Muscle Endurance in Hearing-Impaired Children
Brief Title: Core Stabilization Training on Chest Expansion, Functional Capacity, Trunk Muscle Endurance in Hearing-Impaired Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Assistant professor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/001-002
Record Dates: First submitted 2024-03-29; First posted 2024-04-09 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Core Stabilization; Respiration; Functional Capacity; Endurance; Hearing Impaired Children
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Isometric exercises of the abdominal muscles in the supine, prone, and squatting positions; isotonic exercises in the supine, prone, squatting, and side-lying positions; isotonic exercises in coordination with the extremity movements in the supine, prone, and crawling positions; and trunk rotation exercises in the sitting position will be performed. The Swiss ball will be used for dynamic exercises. It will include isometric and isotonic exercises of the abdominal muscles. Exercises will start with 3 sets of 20 repetitions, gradually increase in intensity on static and dynamic surfaces, and progress towards difficulty. Each exercise will be performed in coordination with breathing control.Breathing control will be coordinated with every exercise.
  Interventions: Other: Core stabilization training
- Control group (No Intervention): Since no training will be given to the control group during the study, we consider it ethically necessary to provide the same training to the control group if it proves effective after the study is over.

INTERVENTIONS:
Other: Core stabilization training — Isometric exercises of the abdominal muscles in the supine, prone, and squatting positions; isotonic exercises in the supine, prone, squatting, and side-lying positions; isotonic exercises in coordination with the extremity movements in the supine, prone, and crawling positions; and trunk rotation exercises in the sitting position will be performed. The Swiss ball will be used for dynamic exercises. It will include isometric and isotonic exercises of the abdominal muscles. Exercises will start with 3 sets of 20 repetitions, gradually increase in intensity on static and dynamic surfaces, and progress towards difficulty. Each exercise will be performed in coordination with breathing control. Breathing control will be coordinated with every exercise.
  Arms: Study group

SUMMARY:
Children's motor skills and physical performance increase with age due to the development of neuromuscular and cardiorespiratory systems. Sensory impairment seen in children with hearing loss can cause balance and coordination disorders, as well as decreased muscle strength and respiratory functions.

Anatomically, core stabilization is provided by the diaphragm, abdominal, hip, pelvic floor, and gluteal muscles. Training for these muscles is intended to improve strength, endurance, and neuromuscular control. This training can help to improve the control of intra-abdominal pressure, intersegmental control of the spine, and muscular control of trunk movement. It also helps in strengthening the respiratory muscles, especially the main inspiratory muscle, the diaphragm. In this study, the effects of core stabilization training on children with hearing impairments' thoracic mobility, functional ability, and trunk muscle endurance will be examined.

DETAILED DESCRIPTION:
Children's motor skills and physical performance increase with age due to the development of neuromuscular and cardiorespiratory systems. Children with hearing loss can display impaired balance and coordination, as well as decreased muscle strength and respiratory functions. Thoracic mobility relates to the function of respiratory muscles that help expand and contract the ribcage. Exercise capacity, or functional capacity, refers to the individual's ability to perform submaximal activities that require the pulmonary, cardiovascular, and skeletal muscle systems to work together and be healthy. Chest wall expansion determines lung volume and functional capacity. A study in patients with chronic obstructive pulmonary disease showed that lung function was positively associated with reduced chest wall expansion.

Core stabilization is provided anatomically by the abdominal muscles in the front, the spinal and gluteal muscles in the back, the diaphragm above, and the pelvic floor and hip muscles below. Core (trunk) stabilization training is a training to increase strength, endurance, and neuromuscular control of the muscles mentioned above. Thus, intersegmental control of the spine, control of intra-abdominal pressure, and muscular control of trunk movement can be improved. It is also beneficial for strengthening the respiratory muscles, especially the diaphragm, which is the main inspiratory muscle.

When the literature was examined, no studies were found that evaluated the effects of exercise on thoracic mobility (chest expansion) and functional capacity in hearing-impaired children. Our planned study is important because it is the first study to evaluate both chest expansion and functional capacity in hearing-impaired children and also because it is the first study to show the effect of the core stabilization exercise program on chest expansion and functional capacity in these children.

ELIGIBILITY:
Inclusion Criteria:

* Presence of clinically diagnosed prelingual sensorineural hearing loss
* Absence of any neurological or orthopedic problems
* Absence of any mental disorder, developmental disorder or syndrome
* Not having participated in any core (trunk) stabilization exercises during the previous six months
* Not having used any medication that would affect respiratory functions in the last 3 months

Exclusion Criteria:

* Intellectual disability that would prevent participation in evaluation and treatment
* Presence of chronic respiratory disease

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Chest expansion | Baseline and immediately after the training
  Chest wall expansion will be measured with a standard measuring tape at three different levels. While the child is in an upright position, with his feet shoulder-width apart and his arms relaxed at his side, measurements will be taken from three areas: at the axilla level (upper level), at the xiphoid level (middle level) and at the subcostal level (lower level).
  The physical therapist standing in front of the child will initially ask the child to breathe normally to determine the tidal volume, after placing the tape measure around the chest. The child will be asked to exhale maximally and then inhale maximally. The difference between the two scales (inhalation - exhalation) will be determined as thoracic expansion (chest expansion). Participants will be instructed to perform three maneuvers and the obtained values will be averaged and recorded. Data will be measured by the same physiotherapist to minimize possible errors due to heterogeneity.

SECONDARY OUTCOMES:
Functional capacity | Baseline and immediately after the training
  The 6-minute walk test (6MWT) is a commonly used submaximal exercise test to assess functional capacity. This test, used to measure cardiovascular endurance, is a clinical indicator of functional capacity and helps measure the ability to perform activities of daily living. The 6MWT will be performed in accordance with The American Thoracic Society guidelines. The participant will be instructed to walk as fast as possible on a 30 m path for 6 minutes, but not to run. The child will sit in a chair close to the starting position and vital values (heart rate and respiratory rate) will be recorded before administering the test. At the end of the test, the distance walked for 6 minutes will be recorded as 6 minutes walking distance (6MWD). After completion of the test, heart rate, respiratory rate will be measured and the child will be asked about the maximum fatigue level after completing the test using the Borg scale.
Trunk muscle endurance | Baseline and immediately after the training
  Curl-up: Measures the muscle endurance of the abdominal muscles. The test begins in a supine position, with the lower extremities abducted at approximately shoulder width and the knees semiflexed. Static back endurance test: Measures the endurance of the back muscles. The test begins in a prone position, with the inguinal area at the end of the table and the pelvis, hips and knees extended flat on the table. Horizontal side bridging: Measures the endurance of the spinal stabilizer muscles. The test begins in a side-lying position with the lower extremities extended and the upper foot placed in front of the lower foot for support.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Tuncer, PhD, PT, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Nuh Naci Yazgan University, Kayseri, Turkey (Türkiye)